CLINICAL TRIAL: NCT06484452
Title: SpO2 Validation Study - Philips FAST 2024
Acronym: FAST 2024
Status: Completed | Type: Observational
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-300177-FAST 2024
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Pulse Oximetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (4):
- Test Group 1: * M1131A (989803205831)
  * M1191T (989803128591)
  * M1191BL (989803144381) for endpoint analysis
  * M1193A (989803205881)
  Interventions: Device: No Intervention
- Test Group 2: * M1194A (989803205891)
  * Alar (989803205381)
  * M1191BL (989803144381) as an internal reference only
  Interventions: Device: No Intervention
- Test Group 3: * EX-Alar on Nasal Ala (Experimental)
  * EX-Alar on Ear (Experimental)
  * M1191BL (989803144381) as an internal reference only
  Interventions: Device: No Intervention
- Test Group 4: * M1133A (989803205851)
  * EX-M1133A (Experimental)
  * M1196T (989803205911)
  * EX-M1196T (Experimental)
  * M1191BL (989803144381) as an internal reference only (optional)
  Interventions: Device: No Intervention

INTERVENTIONS:
Device: No Intervention — No Intervention

SUMMARY:
Validation study to compare the accuracy of non-invasive Philips SpO2 sensors in detecting blood oxygen levels compared to invasive methods requiring a blood draw and lab analysis.

DETAILED DESCRIPTION:
To validate the SpO2 accuracy of the SpO2 sensors under test with the Philips FAST Pulse Oximetry technology during non-motion conditions over the range of 70-100% SaO2, when compared with the reference SaO2 obtained from CO-Oximetry analysis of arterial blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have the ability to understand and provide written informed consent
* Participant is adult between 18-50 years of age
* Participant must be willing and able to comply with study procedures and duration
* Participant is a non-smoker or who has not smoked within 2 days prior to the study.

Exclusion Criteria:

* Participant is considered as being morbidly obese (defined as BMI >39.5)
* Participants with compromised circulation (i.e., Raynaud's Syndrome), injury, or physical malformation of fingers, toes, hands, ears, nose, forehead/skull, or other sensor sites which would limit the ability to test sites needed for the study. Tattoo (e.g. permanent, Henna) or artificial dyes (including spray tan, pigmented tanning lotion) in the optical path which would limit the ability to test sites needed for the study. (Note: Certain malformations may still allow participants to participate if the condition is noted and would not affect the particular sites utilized.)
* Females who are pregnant, who are trying to get pregnant, (confirmed by positive urine pregnancy test unless the participant is known to be not of child-bearing potential)
* Participants who have smoked in the last 2 days or participants who have refrained, for at least 48 hours, with COHb levels >3% as assessed with a Masimo Radical 7 (Rainbow)
* Participants with known respiratory conditions such as: (self-reported)

  * uncontrolled / severe asthma,
  * flu,
  * pneumonia / bronchitis,
  * shortness of breath / respiratory distress,
  * unresolved respiratory or lung surgery,
  * emphysema, COPD, lung disease,
  * Recent COVID (last 2 months)
* Participants with self-reported heart or cardiovascular conditions such as: (self-reported, except for blood pressure and ECG review)

  * high blood pressure: systolic >140 mmHg or diastolic >90 mmHg on 3 consecutive readings (reviewed during health screen),
  * have had cardiovascular surgery, except successful minor surgery without clinical symptoms (i.e., PFO, PDA),
  * chest pain (angina),
  * heart rhythms other than a normal sinus rhythm or with respiratory sinus arrhythmia (reviewed during health screen),
  * previous heart attack,
  * blocked artery,
  * unexplained shortness of breath,
  * congestive heart failure (CHF),
  * history of stroke,
  * transient ischemic attack,
  * carotid artery disease,
  * myocardial ischemia,
  * myocardial infarction,
  * cardiomyopathy,
  * implantable active medical device such as pacemaker or automatic defibrillator
* Participants with self-reported health conditions as identified in the Health Assessment Form

  * diabetes,
  * uncontrolled thyroid disease,
  * kidney disease / chronic renal impairment,
  * history of seizures (except childhood febrile seizures),
  * epilepsy,
  * history of unexplained syncope,
  * recent history of frequent migraine headaches,
  * recent symptomatic head injury (within the last 2 months),
  * Cancer requiring chemotherapy, radiation, or current treatment
* Participants with known clotting disorders (self-reported)

  * history of bleeding disorders or personal history of prolonged bleeding from injury,
  * history of blood clots,
  * hemophilia,
  * current use of blood thinner: prescription or daily use of aspirin,
  * Sickle Cell Trait or Disease
* Participants with self-reported dermatological conditions at sensor application sites
* Severe dermatitis,
* Hyperkeratosis,
* Nail fungus
* Participants with severe contact allergies to standard adhesives, latex, silicone or other materials found in pulse oximetry sensors, ECG electrodes, respiration monitor electrodes or other medical sensors (self-reported)
* Participants with severe allergies to iodine (only applicable if iodine is used)
* Participants with severe allergies to lidocaine (or similar pharmacological agents, e.g. Novocaine),
* Failure of the Perfusion Index Ulnar/Ulnar+Radial Ratio test (Ratio <0.4)
* Unwillingness or inability to remove colored nail polish or artificial nails from test digits
* Participants with stretched or dilated piercings at the application site of ear sensors. (Applicable for test groups with M1194A and EX-Alar on ear only.)
* Participant received intravascular dye within the past 48 hours (e.g. Indocyanine green, methylene blue, dyes used in cardiac output monitoring)
* Surgical hardware in pathway of Device Under Test
* Other known health condition, should be considered upon disclosure in health assessment form

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population for this protocol will include a minimum of 96 to a maximum of 120 healthy, competent adult male and female participants of any race and ranging in pigmentation from light to dark. Participants will be non-smoking (or have refrained from smoking for 2 days) and between the ages of 18-50 years old.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-08-29 (Actual)

PRIMARY OUTCOMES:
SpO2 Accuracy | May-August 2024
  Accuracy expressed in ARMS of SpO2 measurements obtained from the SpO2 sensors under test with the Philips Pulse Oximetry technology over the range of 70-100% SaO2, in comparision to SaO2 as ground truth.

SECONDARY OUTCOMES:
Non-Disparate Bias | May-August 2024
  Non-disparate bias and differential mean bias of the SpO2 sensors under test in the SaO2 ranges of 70% ≤ SaO2 ≤ 85% and 85% < SaO2 ≤ 100%.

CONTACTS AND LOCATIONS:
Locations (1):
- Element Materials Technology, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Study did NOT meet the ACT requirments and will not have results posted.